CLINICAL TRIAL: NCT01794728
Title: How the Elderly Live With Pain in Heart Failure
Acronym: HELP-HF
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12D.115
Record Dates: First submitted 2012-12-21; First posted 2013-02-20 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure
Keywords: Pain Management
MeSH Terms: conditions — Heart Failure; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly inpatients with heart failure: A single cohort group of elderly patients hospitalized for heart failure.

SUMMARY:
The How the Elderly Live with Pain in Heart Failure (HELP-HF) study provides the opportunity to assess the complaints of pain in a cohort of HF patient admitted to Thomas Jefferson University Hospital (TJUH). Additional information on their existing co-morbid conditions, an inventory of their prescribed medications, and details regarding the type of treatment interventions (over the counter analgesia and other comfort practices) they report using will be collected.

DETAILED DESCRIPTION:
Study Events Patients admitted to TJUH with a HF diagnosis will be identified by intensive clinical research coordinator screening methods. The potential subjects will be approached in the acute care area for interview and consent to participate. At that visit, the variables of interest will be collected and the questionnaires completed. Following discharge, the subjects will be re-interviewed at follow-up clinic visits or by telephone, depending on whether the visit is to a Jefferson University Physician provider or to an outside provider or as circumstances allow.

Subjects will sign an informed consent to participate in HELP-HF. A selection of assessment questionnaires (listed below) and performance measures will be completed during the index hospitalization and at a subsequent follow up clinic visits or by telephone call. Some of these assessments involve data collection from standard of care encounters or tests and will be abstracted from the medical record.

The Kansas City Cardiomyopathy Questionnaire (KCCQ) The KCCQ is a valid, reliable and responsive health status measure for HF patients and serves as a clinically meaningful outcome assessment tool that is widely used in cardiovascular research, patient management, and quality of life self-assessment.12 The Brief Pain Inventory (BPI) The BPI is one of the most widely used measurement tools for assessing clinical pain. It allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. Initially developed to assess pain related to cancer, the BPI has validated as an appropriate measure for pain caused by a wide range of clinical conditions. , The Charlson Co-Morbidity Index (CCI) Comorbidity describes the effect of all other diseases an individual patient might have other than the primary disease of interest. The CCI is used to characterize comorbid medical conditions and allows inferences about the extent to which symptoms and other factors related to quality of life may be attributable to conditions other than HF. The CCI designates comorbid conditions in 19 categories and each category has an associated weight based on the adjusted risk of one-year mortality, and the overall comorbidity score reflects the cumulative increased likelihood of one-year mortality. Charlson scores can range between 0 and 35, with a higher score indicating increase in burden of comorbid disease.

OTC Medication Inventory A comprehensive list of any over the counter (OTC) medications will be collected and reconciled via review of the electronic medical records and by subject interview.

Brief Interventions Measures (BIM) The BIM questionnaire is a novel tool developed for use in the HELP-HF study. It is adapted from similar questionnaires used in palliative oncology care and incorporates an inventory of comfort measure identified in the literature. These include measures like application of heat or cold, massage, and other self-selected therapies.

Case Report Form and Data Capture A paper case report form (data collection tool) will be developed for each subject's study records. All data will be entered by study personnel into a password-protected database using the REDCap (Research Electronic Data Capture) system. REDCap is a secure, web-based application designed to support electronic data capture for research studies. REDCap is used by selected areas within the University. It is a service available via a free collaboration with the NIH CTSA structure and accessed at TJU with permission and oversight via internal Information Systems at the University's Kimmel Cancer Center. REDCap allows for monitored dual data entry via a web-based system that is maintained on a protected server and will be used by the study investigators, coordinators and statistician.

Statistical Analyses Plan Subject demographics and co-morbidities as well as characteristics of the self-reported pain, treatment selections, and efficacy will be reported as medians and interquartile ranges (IQRs) for continuous variables and as percentages of non-missing values for categorical variables. Patients will be stratified by pain scores. Univariate comparisons between patients with and without pain will be performed using the Pearson χ2 test for categorical variables and the Wilcoxon rank-sum test for continuous and ordinal variables.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 60 years.
* Admission to hospital for worsening HF

Exclusion Criteria:

* History of uncontrolled hypertension.
* Severe valve disease.
* End-stage (Stage D) HF, including treatment with chronic ionotropic drugs or left ventricular assist device support.
* Advanced malignancy or other medical condition with life expectancy less than 2 years or undergoing active chemotherapy or radiation therapy.
* Advanced chronic kidney disease (CKD) defined as estimated glomerular filtration rate (GFR) < 20 mL/min/1.73 m2 based upon the Modification of Diet in Renal Disease (MDRD) study equation), or on chronic or intermittent dialysis or dialysis anticipated within the next 6 months.
* Chronic anemia with hemoglobin < 9 gm/dl for males, < 8 gm/dl for females or acute anemia requiring transfusion of 2 or more units of blood.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women age 60 or greater hospitalized with acute decompensated heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in characteristics and frequency of pain in a cohort of HF patients | Time of enrollment date and after 30 days.
  Assessment will be completed at baseline time of enrollment during hospitalization and again at 30 days after discharge. The instrument used is the Brief Pain Inventory questionnaire.

SECONDARY OUTCOMES:
Change in the analgesia and comfort measures selected to treat pain by a cohort of HF patients | Time of enrollment date and after 30 days.
  Assessment will be completed at baseline time of enrollment during hospitalization and again at 30 days after discharge. The instrument used is a modified Pain Intervention Measurement questionnaire.
Change in the relationship between pain and self- reported QOL in a cohort of HF patients | Time of enrollment date and after 30 days.
  Assessment will be completed at baseline time of enrollment during hospitalization and again at 30 days after discharge. The instrument used is the Kansas City Cardiomyopathy questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David J Whellan, MD MHS, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States